CLINICAL TRIAL: NCT00359138
Title: A Double-blind, Double-dummy, Parallel-group, Placebo-controlled, Randomized Study to Assess the Duration of the Suppressive Effects of Desloratadine on the Cutaneous Allergen-induced Wheal and Flare (1) Response After Discontinuation
Brief Title: The Duration of the Suppressive Effects of Desloratadine on Allergen Prick Tests After Discontinuation (P04441)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04441
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypersensitivity
Keywords: Histamine H1 Antagonists; Anti-Allergic Agents
MeSH Terms: conditions — Hypersensitivity | interventions — desloratadine; levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desloratadine 5 mg tablet + Levocetirizine placebo capsule (Experimental): Subject was instructed to take 1 tablet and 1 capsule, once daily from day one (visit 3) to day 8 (visit 4).
  Interventions: Drug: desloratadine; Drug: Levocetirizine placebo capsule
- Desloratadine placebo tablet + Levocetirizine 5 mg capsule (Active Comparator): Subject was instructed to take 1 tablet and 1 capsule, once daily from day one (visit 3) to day 8 (visit 4).
  Interventions: Drug: levocetirizine; Drug: Desloratadine placebo tablet
- Desloratadine placebo tablet + Levocetirizine placebo capsule (Placebo Comparator): Subject was instructed to take 1 tablet and 1 capsule, once daily from day one (visit 3) to day 8 (visit 4).
  Interventions: Drug: Desloratadine placebo tablet; Drug: Levocetirizine placebo capsule

INTERVENTIONS:
Drug: desloratadine — 5 mg tablet once daily
  Arms: Desloratadine 5 mg tablet + Levocetirizine placebo capsule
Drug: levocetirizine — 5 mg capsule once daily
  Arms: Desloratadine placebo tablet + Levocetirizine 5 mg capsule
Drug: Desloratadine placebo tablet — once daily
  Arms: Desloratadine placebo tablet + Levocetirizine 5 mg capsule; Desloratadine placebo tablet + Levocetirizine placebo capsule
Drug: Levocetirizine placebo capsule — once daily
  Arms: Desloratadine 5 mg tablet + Levocetirizine placebo capsule; Desloratadine placebo tablet + Levocetirizine placebo capsule

SUMMARY:
This is a randomized, double-blind, double-dummy, placebo-controlled, parallel-group, single center study in subjects with positive histamine skin prick test and a positive RadioAllergoSorbent Test (RAST) (class > 2) to one of the tested standardized allergenic extracts: tree pollen, cat dander, house dust mite, or a mixture of five grass pollens. Subjects will be randomized to desloratadine 5 mg once daily, levocetirizine 5mg once daily, or placebo once daily for 8 days of treatment followed by 11 days of skin testing after discontinuation of the antihistamine treatment phase. The duration of the suppressive effects of desloratadine on cutaneous allergen-induced wheal and flare responses after discontinuation of a one-week treatment will be established.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older, of either sex.
* Subjects must have at least a history of positive skin testing to the allergens of tree pollen, grass pollen, house dust mite, or cat dander.
* Non symptomatic volunteers allergic of different pollen they must be included out of the specific pollinic season.
* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must understand and be able to adhere to visit schedules
* Subjects must be in general good health.
* Women of child-bearing potential must have a negative pregnancy test at Day -1 and must use an accepted method of contraception during the entire duration of the study.

Exclusion Criteria:

* Subjects who have persistent asthma.
* Subjects who have chronic urticaria or atopic dermatosis.
* Subjects who have received any treatment listed below more recently than the indicated washout period prior to Randomization, or who must continue to receive treatment as listed below.

Medications Prohibited During the Trial and Washout Period Prior to Visit 1

* Corticosteroids

  * Intramuscular or intra-articular, 1 month
  * Oral, inhaled, intravenous, rectal, intranasal, or ocular, 7 days
  * High-potency dermatological, 7 days
* Cromolyn/Lodoxamide/Nedocromil

  * Intranasal, ocular, inhaled, or oral, 2 days
* Antihistamines

  * Long-acting prescription (eg, levocetirizine, fexofenadine, and desloratadine), 15 days
  * Short-acting (eg, chlorpheniramine, brompheniramine including over-the-counter [OTC] forms, hydroxyzine), 15 days
  * Ocular (eg, levocabastine), 15 days
* Leukotriene inhibitors (eg, montelukast), 7 days
* Systemic antibiotics, 14 days (the washout refers to antibiotics used to treat an upper or lower respiratory tract infection)
* Immunotherapy (desensitization), 1 year
* Decongestants

  * oral, 2 days
  * local, 2 days
* Ophthalmic non-steroidal anti-inflammatory drugs (NSAIDs; eg, Toradol), 5 days
* Investigational medications, 30 days
* Tricyclic antidepressants (eg, amitriptyline, clomipramine, doxepin, imipramine, trimipramine, amoxapine, desipramine, nortriptyline, protriptyline), 30 days
* Tetracyclic antidepressants (eg, maprotiline, mirtazapine), 30 days

  * Subjects with a history of hypersensitivity to desloratadine, to levocetirizine, or any of their excipients.
  * Women who are breast-feeding, pregnant, or intend to become pregnant.
  * Subjects with any clinically significant condition or situation, other than the condition being studied, that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study.
  * Subjects who have used any investigational drugs within 30 days of randomization.
  * Subjects working between 11 PM and 8 AM (night shift).
  * Subjects who have skin/color pigmentation incompatible with accurate measurements of flare reaction.
  * Subjects with cutaneous hyperactivity: negative prick test control >3 mm.
  * Subjects who are participating in any other clinical study.
  * Subjects who are part of the staff personnel directly involved with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Desloratadine 5 mg Tablet + Levocetirizine Placebo Capsule | Desloratadine Placebo Tablet + Levocetirizine 5 mg Capsule | Desloratadine Placebo Tablet + Levocetirizine Placebo Capsule
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desloratadine 5 mg Tablet + Levocetirizine Placebo Capsule | Desloratadine Placebo Tablet + Levocetirizine 5 mg Capsule | Desloratadine Placebo Tablet + Levocetirizine Placebo Capsule | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.42 (4.91) | 28.33 (8.69) | 28.83 (11.55) | 26.86 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 5 | 18
  Male | 7 | 4 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Duration of Suppressive Effect of Desloratadine After Discontinuation of a 1-week Treatment
Description: The number of days after treatment discontinuation until a measurable wheal and flare response.
Time Frame: Starting at Day 8
Measure: Mean (Standard Error); unit: Days
Arm/Group | Desloratadine 5 mg Tablet + Levocetirizine Placebo Capsule | Desloratadine Placebo Tablet + Levocetirizine 5 mg Capsule | Desloratadine Placebo Tablet + Levocetirizine Placebo Capsule
Number analyzed (Participants) | 12 | 12 | 12
Days | 5 (1.65) [0.4613 to 0.9400] | 4 (1.60) | NA (NA) — Results are based on the individual active group relative to placebo. Not applicable for placebo relative to placebo

ADVERSE EVENTS:
Arm/Group | Desloratadine 5 mg Tablet + Levocetirizine Placebo Capsule | Desloratadine Placebo Tablet + Levocetirizine 5 mg Capsule | Desloratadine Placebo Tablet + Levocetirizine Placebo Capsule
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 4/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desloratadine 5 mg Tablet + Levocetirizine Placebo Capsule (N=12) | Desloratadine Placebo Tablet + Levocetirizine 5 mg Capsule (N=12) | Desloratadine Placebo Tablet + Levocetirizine Placebo Capsule (N=12)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less